CLINICAL TRIAL: NCT07403513
Title: The Role of Climate Change Education on Awareness, Concern, and Hope in Pregnant Women: A Randomized Controlled Trial
Brief Title: The Role of Climate Change Education on Awareness, Concern, and Hope in Pregnant Women
Acronym: Climate Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Sevilay Aydın Çelik, Specialist Nurse, PhD Student, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SBU-SBE-SAC-02
Record Dates: First submitted 2026-01-29; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Climate Change; Pregnancy
Keywords: climate change; pregnancy; mother health; health education; anxiety; hope
MeSH Terms: conditions — Health Education; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Climate Change Education Intervention Group (Experimental): The initiative group, consisting of 77 participants, will receive approximately 60 minutes of in-person training on "Pregnancy and Climate Change" following a pre-test. The training will cover environmental risk factors, their effects on pregnancy, methods of contraception, and individual awareness; informative brochures will be distributed to participants after the training. The final test data for the initiative group will be collected four weeks after the training.
  Interventions: Other: Climate Change Education
- Control Group (No Climate Change Education) (No Intervention): The control group, consisting of 77 participants, will receive only a pre-test and a post-test four weeks later, without any training.

INTERVENTIONS:
Other: Climate Change Education — The intervention group will receive approximately 60 minutes of in-person training on "Pregnancy and Climate Change" following the pre-test. The training will focus on environmental risks, their effects on pregnancy, and contraceptive approaches; an informative brochure will be provided at the end of the training. The final test measurements for the intervention group will be taken four weeks after the training.
  Arms: Climate Change Education Intervention Group

SUMMARY:
Climate change can negatively impact women's health at different stages of life through environmental risks such as extreme temperatures, vector-borne diseases, and air pollution. Particularly during pregnancy, a period of intense physiological and psychosocial changes, climate change is reported to be associated with adverse maternal and infant outcomes such as spontaneous abortion, preterm birth, low birth weight, intrauterine growth retardation, and neonatal mortality. Therefore, identifying climate change-related risks during pregnancy, raising awareness of these risks, and developing preventative approaches are crucial for protecting maternal and fetal health.

This study aims to evaluate the impact of a "Pregnancy and Climate Change" education program developed for pregnant women on their climate change awareness levels, anxiety levels regarding climate change, and hope levels for preventing climate change. The effectiveness of the education program will be determined by comparing the pre-test and post-test scores of the intervention and control groups.

The research is designed as a randomized controlled experimental study with experimental and control groups in a pre-test-post-test configuration. The study population consists of all pregnant women who applied to the antenatal outpatient clinic of Zeynep Kamil Women and Children's Diseases Training and Research Hospital. The sample will consist of pregnant women who are 18 years of age and older, have a gestational age of 32 weeks or less, can speak and understand Turkish, and volunteer to participate in the study. Pregnant women with a history of psychiatric illness, systemic disease before or during pregnancy, or who experienced pregnancy complications such as preeclampsia and gestational diabetes will be excluded from the study.

The sample size was calculated using the G*Power 3.1 program based on the independent samples t-test. A moderate effect size (Cohen's d = 0.50), a 95% confidence level, and 80% statistical power were used. The analysis determined that a total of 128 pregnant women were needed, with at least 64 participants in each group. Considering possible sample losses, a 20% increase was made, and the study was planned with a total of 154 pregnant women, with 77 pregnant women in each group. Participants will be assigned to intervention (n=77) and control (n=77) groups using computer-assisted block randomization.

The intervention group will receive approximately 60 minutes of face-to-face training on "Pregnancy and Climate Change" following a pre-test. The training will cover environmental risk factors, their effects on pregnancy, individual contraceptive approaches, and information aimed at raising awareness. Informative brochures will be distributed to participants after the training. Post-test data for the intervention group will be collected four weeks after the training. The control group will receive only a pre-test and a post-test four weeks later, without any training.

Data will be collected through face-to-face interviews using a Personal Information Form, the Climate Change Anxiety Scale, the Climate Change Awareness Scale, and the Hope Scale for Preventing Climate Change. Data analysis will be performed using SPSS 25.0 software; descriptive statistics, t-test, ANOVA, chi-square test, and normal distribution analysis will be utilized.

DETAILED DESCRIPTION:
Climate change-related problems such as extreme heat, vector-borne diseases, and air pollution can negatively affect women's health at different stages of life. Pregnancy is a period characterized by significant physiological and psychosocial changes, during which women may be particularly vulnerable to environmental stressors. During this period, exposure to the effects of climate change has been associated with adverse maternal and fetal outcomes, including spontaneous abortion, preterm labor, low birth weight, intrauterine growth retardation, and neonatal mortality. Identifying climate change-related risks during pregnancy, increasing awareness of these risks, taking preventive measures, and minimizing negative outcomes after problems occur are essential for protecting and improving maternal and fetal health.

Research Objectives

The objectives of this study are:

To evaluate the effect of a "Pregnancy and Climate Change" education program on pregnant women's levels of climate change awareness,

To determine the effect of the education program on pregnant women's anxiety related to climate change,

To examine the effect of the education program on pregnant women's hope levels regarding the prevention of climate change, and

To assess the effectiveness of the education program by comparing pre-test and post-test scores between the intervention and control groups.

Research Design

This study is planned as a randomized controlled experimental study with a pre-test-post-test design, including an intervention group and a control group.

Research Population and Sample

The research population consists of all pregnant women who apply to the maternity clinic of Zeynep Kâmil Women and Children's Diseases Training and Research Hospital. Pregnant women who meet the inclusion criteria will be included in the study.

The inclusion criteria are as follows: being 18 years of age or older, being at or below 32 weeks of gestation, being able to speak and understand Turkish, and volunteering to participate in the study. Pregnant women with a history of psychiatric illness or psychiatric treatment, those with systemic diseases before or during pregnancy, or those who have experienced pregnancy-related complications such as preeclampsia or gestational diabetes will be excluded from the study.

Sample Size

The sample size was calculated using a power analysis based on an independent samples t-test. A moderate effect size, a significance level of 0.05, and a statistical power of 0.80 were used. Based on these parameters, a minimum of 128 participants was required, with at least 64 participants in each group. Considering possible sample loss, the sample size was increased by 20%, and the study was planned to be conducted with a total of 154 pregnant women, with 77 participants in the intervention group and 77 participants in the control group.

Randomization and Intervention

Participants will be assigned to the intervention and control groups using computer-assisted block randomization. The randomization process will be carried out by a research assistant independent of the researcher to ensure allocation concealment.

Participants in the intervention group will receive approximately 60 minutes of face-to-face training on "Pregnancy and Climate Change" after completing the pre-test. The training content will include environmental risk factors, the effects of climate change on pregnancy, individual protective measures, and awareness-raising strategies. At the end of the training session, participants will be provided with an informational brochure summarizing the key topics. Post-test data for the intervention group will be collected four weeks after the training.

Participants in the control group will receive only the pre-test and will not receive any training. Post-test data for the control group will also be collected four weeks after the pre-test. Data collection will therefore be conducted simultaneously in both groups to ensure comparability.

Data Collection Tools

Data will be collected through face-to-face interviews using a personal information form and standardized measurement tools assessing climate change awareness, climate change-related anxiety, and hope related to preventing climate change. The personal information form includes questions on sociodemographic characteristics, general health status, and obstetric history.

Ethical Considerations

Prior to data collection, ethical approval will be obtained from the Ethics Committee of Zeynep Kâmil Women and Children's Diseases Training and Research Hospital, and institutional permission will be obtained from the hospital administration. Participants will be informed that their participation is voluntary, their personal information will remain confidential, the data will be used only for scientific purposes, and they may withdraw from the study at any time without consequences. The study will begin only after obtaining both verbal and written informed consent from all participants.

Limitations

The main limitation of this study is that it will be conducted in a single center with a limited sample size.

Data Analysis

All collected data will be transferred to a computer environment and checked for accuracy and completeness. Statistical analyses will be performed using a statistical software package. Descriptive statistics such as mean, standard deviation, minimum, maximum, frequency, and percentage will be calculated. Normality of the data will be assessed using appropriate distribution tests. Group comparisons will be performed using parametric statistical tests, and categorical variables will be analyzed using chi-square tests. Statistical significance will be evaluated at a 0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* Being pregnant
* Being 18 years of age or older
* Being at or below 32 weeks of gestation
* Ability to speak and understand Turkish
* Volunteering to participate in the study

Exclusion Criteria:

* History of psychiatric illness or psychiatric treatment
* Presence of any systemic disease before or during pregnancy
* History of pregnancy-related complications, such as preeclampsia or gestational diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant Women
Enrollment: 154 (Actual)
Dates: Start 2025-07-09 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Climate Change Awareness Scale | 6 Month
  Assesses participants' knowledge and understanding of climate change, environmental risks, and preventive behaviors. Measured using the Climate Change Awareness Scale (CCAS) at baseline and four weeks after the intervention.High scores on the scale indicate high awareness.

SECONDARY OUTCOMES:
Climate Change Anxiety Scale | 6 Month
  Evaluates participants' levels of anxiety and perceived helplessness related to climate change. Assessed with the Climate Change Concern Scale (CCCS) at baseline and post-intervention. Higher scores indicate greater concern.

OTHER OUTCOMES:
Hope for Climate Change Prevention Scale | 6 Month
  Measures participants' sense of hope and perceived ability to prevent climate change. Assessed using the Hope for Climate Change Prevention Scale (HCCPS) before and four weeks after the intervention. Higher scores indicate greater hope.

CONTACTS AND LOCATIONS:
Overall Officials: Melike DİŞSİZ, Associate Professor, PhD RN, Principal Investigator — Istanbul Health Sciences University Hamidiye Faculty of Nursing
Locations (1):
- Istanbul Health Sciences University Hamidiye Institute of Health Sciences, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be shared in a fully de-identified and anonymized format. Shared data will be used solely for scientific research purposes and cannot be linked to identifiable participants. Data will be made available upon request, following appropriate ethical and legal approvals.